CLINICAL TRIAL: NCT06233292
Title: A Phase 1/2 Dose Escalation, Tolerability, Safety and Pharmacokinetics Study of ZG005 in Patients With Advanced Solid Tumors
Brief Title: A Study of ZG005 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-001
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): The study will begin with open-label dose escalation in ZG005 monotherapy treatment to determine the Maximum tolerated dose (MTD).
  Interventions: Biological: ZG005 Powder for Injection
- Part 2: Dose Expansion: Recommended Phase 2 Dose (RP2D) of ZG005 monotherapy (Experimental): The dose-expansion stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage.Single drug dose expansion was performed in different tumors, such as :Non-small cell lung cancer, small cell lung cancer, Esophageal squamous cell carcinoma, Alveolar soft part sarcoma
  Interventions: Biological: ZG005 Powder for Injection

INTERVENTIONS:
Biological: ZG005 Powder for Injection — The dose groups of ZG005 for dose escalations are set as 0.3 mg/kg, 1mg/kg, 3mg/kg, 10mg/kg, and 20mg/kg, intravenous infusion, once every 3 weeks.
  Other Names: ZG005
  Arms: Part 1: Dose Escalation
Biological: ZG005 Powder for Injection — Recommended Phase 2 Dose (RP2D) of ZG005 monotherapy, intravenous infusion, once every 3 weeks.
  Other Names: ZG005
  Arms: Part 2: Dose Expansion: Recommended Phase 2 Dose (RP2D) of ZG005 monotherapy

SUMMARY:
This is a multi-center, open-label, Phase 1/2 study of ZG005 for the treatment of subjects with advanced solid tumors, and consists of three stages: dose escalation and confirmation of MTD/recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-70 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
* Life expectancy ≥ 3 months;
* Histologically or cytologically confirmed diagnosis of advanced solid tumors.

Exclusion Criteria:

* Medical history, computed tomography (CT) or magnetic resonance imaging (MRI) results indicate that existence of the central nervous system(CNS) metastases;
* Any other malignancy within 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 21Days
  A DLT is defined as any of the following ≥ Grade 3 adverse events occurring from the first dose to the end of first Cycle (21 days), unless the investigator deems that the AE is clearly related to the disease progress or definitely due to an external cause.
Adverse Event (AE) | Up to 24 Months
  Number of participants with adverse events that are related to treatment
Objective Response Rate | Up to 24 Months
  Objective response rate was based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Maximum tolerated dose (MTD) | Up to 24 Months
  During the dose escalation stage, if 2 of up to 6 subjects in the first dose groups experienced DLT, then the dose level will be considered to be an intolerable dose or DLT dose level, and the previous lower dose will be considered to be the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No